CLINICAL TRIAL: NCT01631929
Title: Two Bag System vs. One Bag System for Hydration Patients With Diabetic Ketoacidosis
Brief Title: Two Bag System for Hydration in Diabetes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Monitoring Committee found significant & meaningful difference on main outcome
Sponsor: Hospital General de Niños Pedro de Elizalde (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 65-HGNPE-2012
Record Dates: First submitted 2012-06-25; First posted 2012-06-29 (Estimated); Results first posted 2015-10-26 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2016-12

CONDITIONS: Diabetes; Ketoacidosis
Keywords: Diabetes; Ketoacidosis; Children
MeSH Terms: conditions — Diabetes Mellitus; Ketosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- One bag (Active Comparator): IV infusion of fluids, electrolytes and dextrose using one bag
  Interventions: Other: One bag
- Two bags (Experimental): Using 2 bags with different solutions with the same electrolyte content but different dextrose concentration (0% and 10%), administered simultaneously through the same intravenous line.
  Interventions: Other: Two bags

INTERVENTIONS:
Other: One bag — Infusion of dextrose and electrolytes using one bag
  Arms: One bag
Other: Two bags — Using 2 bags with different solutions with the same electrolyte content but different dextrose concentration (0% and 10%), administered simultaneously through the same intravenous line.
  Arms: Two bags

SUMMARY:
This is a randomized controlled trial comparing the time needed to get the conditions to space hourly controls to controls every 4 hours, using the one bag system versus the two bags system, in the initial treatment of children with diabetic ketoacidosis. After fast infusion of isotonic saline solution (20 ml/kg) to prevent shock, the administration of maintenance fluids and insulin therapy is indicated. Hourly plasmatic levels of glucose controls could determine changes in glucose IV administration. On using the classic one bag system each change determine a bag change. Using the two bag system allows to deliver the patient the appropriate glucose infusion in less time.

DETAILED DESCRIPTION:
The treatment of children with diabetic ketoacidosis includes fast infusion of isotonic saline solution to prevent shock (20 ml/kg), and then the administration of maintenance fluids and insulin therapy according to hourly plasmatic glucose levels controls. Finally, after patients stabilization, controls becomes less frequents (each 4 hours).

During the stabilization period infusion of glucose is calculated hourly according to plasmatic glucose levels. These modifications in IV infusion can be very frequent, sometimes by the hour, requiring preparation of a new solution for hydration (in a new bag).

This procedure takes time, during which the patient continues receiving the previous IV infusion until the changes are effectively made. Therefore, usually changes are not strictly hourly, interfering with the adjustment of the organism to the above mentioned changes.

The 2 bag system consists in using 2 bags with different solutions with the same electrolyte content but different dextrose concentration (0% and 10%), administered simultaneously through the same intravenous line. Using this system allows that changes needed in the administration of fluids and/or dextrose, may be easily and instantly managed by delivering different amounts from each bag to achieve the desired infusion rate without having to replace the bag.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 1 to 18 years old
* Diabetic ketoacidosis(plasmatic glucose > 250mg/dl, pH < 7.3, bicarbonate < 15mmol/L, ketonuria and glycosuria)

Exclusion Criteria:

* Patients who already received insulin in the Emergency Department.
* Patients who, because of their clinical condition, require admission to intensive care unit.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2012-08; Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan P Ferrira, MD, Principal Investigator — Hospital General de Niños Pedro de Elizalde
Locations (1):
- Hospital General de NIños Pedro de Elizalde, Buenos Aires, Argentina

REFERENCES:
- [Background] Poirier MP, Greer D, Satin-Smith M. A prospective study of the "two-bag system'' in diabetic ketoacidosis management. Clin Pediatr (Phila). 2004 Nov-Dec;43(9):809-13. doi: 10.1177/000992280404300904. PMID 15583776
- [Result] Grimberg A, Cerri RW, Satin-Smith M, Cohen P. The "two bag system" for variable intravenous dextrose and fluid administration: benefits in diabetic ketoacidosis management. J Pediatr. 1999 Mar;134(3):376-8. doi: 10.1016/s0022-3476(99)70469-5. PMID 10064682

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | One Bag | Two Bags
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | One Bag | Two Bags | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 6 | 12
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.83 (1.7) | 9.67 (2.7) | 9.2 (3.4)
Gender [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 1 | 1 | 2
Disease debuted [Number; unit: participants]
  Yes | 4 | 2 | 6
  Not | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Time to Achieve Patient Stabilization
Description: Time needed to achieve patient stabilization defined by:
  * Plasmatic glucose < 250 mg/dl
  * Blood pH > 7.3
  * Plasmatic bicarbonate > 15 mmol/L
Time Frame: Participants were followed for the duration of ketoacidosis (an expected average of 12 hours)
Measure: Mean (95% Confidence Interval); unit: Hours
Arm/Group | One Bag | Two Bags
Number analyzed (Participants) | 6 | 6
Hours | 13.3 [10.5 to 16.1] | 9.8 [8.64 to 10.96]

ADVERSE EVENTS:
Arm/Group | One Bag | Two Bags
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No